CLINICAL TRIAL: NCT04049955
Title: Endoscopic Management of Fistulas Related to Sleeve Gastrectomy With Double Pigtail Stents According to the BARTOLI Technique : an Interventional Multicentric and Prospective Study.
Brief Title: Endoscopic Management of Fistulas Related to Sleeve Gastrectomy With Double Pigtail Stents According to the BARTOLI Technique
Acronym: bartoli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Bichat Hospital (Other); centre hospitalier de Compiegne (Unknown); clinique des cedres, Cornebarrieu (Unknown); Centre Hospitalier Universitaire de Nīmes (Other); Centre Hospitalier de Saint-Brieuc (Other); Hospital Prive Jean Mermoz (Other); Centre Hospitalier Universitaire de Nice (Other); Nantes University Hospital (Other); Rennes University Hospital (Other); Centre Hospitalier Toulon (Unknown); Centre Hospitalier Universitaire de Besancon (Other); Clinique Paris-Bercy (Other); University Hospital, Bordeaux (Other); Saint Antoine University Hospital (Other); Hôpital Edouard Herriot (Other); University Hospital, Brest (Other); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0017
Record Dates: First submitted 2019-07-18; First posted 2019-08-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Gastrostomy; Fistula
Keywords: sleeve gastrostomy; endoscopy; fistula; double pig tail stents
MeSH Terms: conditions — Fistula | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopy (Experimental): In the case of a well-organized abscessed collection responsible for sepsis instability, or poorly organized collection, an external drainage is carried out, by a radiological or a surgical way. The endoscopy is performed 7 days later. If there is no hemodynamic instability and in presence of a well-organized abscessed collection, a first-line endoscopy is carried out. After laying 2 double pig tail stents, the external drainage is removed 2 to 7 days later.
  Interventions: Procedure: endoscopy

INTERVENTIONS:
Procedure: endoscopy — In the case of a well-organized abscessed collection responsible for sepsis instability, or poorly organized collection, an external drainage is carried out, by a radiological or a surgical way. The endoscopy is performed 7 days later. If there is no hemodynamic instability and in presence of a well-organized abscessed collection, a first-line endoscopy is carried out. After laying 2 double pig tail stents, the external drainage is removed 2 to 7 days later.

SUMMARY:
Obesity is a major health problem in western countries, and sleeve gastrectomy has proven its effectiveness on weight loss and improvement of comorbidities related to obesity. The main complication is the occurrence of upper fistula (2%), and may be responsible of several deaths.

There is no consensus on medical, radiological and surgical management of fistula. It depends on the resources of each center and is based on a low level evidence The inconstant efficacy of the endoscopic treatment by closing fistula (digestive stents, clips, glue) motivates a new endoscopic approach. It consists of an internal drainage of the collection by using double pigtail stents through the fistulous orifice.

DETAILED DESCRIPTION:
Partially or fully covered stents are the most used method, but are not supported by any comparative studies. Their results are inconstant and the closure rate is estimated between 15 and 100%, with a hazardous median healing time. This method is associated with frequent complications, such as spontaneous migrations, impactions or ulcerations responsible for potentially fatal hematemesis. The preliminary results of using OTSC clips (OVESCO®) seem encouraging, but this technique requires external drainage to obtain a collection free from infection. A new approach is to perform an internal drainage of the peri-orificial collection by using double pigtail stents through the fistulous orifice and to direct the fistula closure from the outside to the inside. This endoscopic treatment, combined with nutritional support and initial antibiotic therapy, allows rapid weaning of external drainage and short healing times. CT and endoscopic evaluation are needed at the sixth week for stents removal in the event of a favorable evolution. In the opposite case, a second endoscopic treatment is performed. In case of unfavorable evolution, a radical surgical treatment, in the absence of endoscopic alternative, will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Any major patient hospitalized for a symptomatic fistula after sleeve gastrectomy, outside the exclusion criteria, is eligible.
* Free, informed and signed consent
* Affiliation to the social security system

Exclusion Criteria:

* Other surgery than Sleeve gastrectomy
* Fistula located at a site other than the upper pole of the staple line
* Fistulization on the upper diaphragmatic floor
* Fistulous orifice larger than 25 mm
* Pregnancy
* Patient under guardianship or curators or deprived of public law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Fistula Healing at week 18 | week 18 after endoscopy
  Number of Participants with Healing at week 18

SECONDARY OUTCOMES:
Number of Participants with Fistula Healing at week 6 | week 6 after endoscopy
  Number of Participants with Fistula Healing at week 6
Number of Participants with Fistula Healing at week 12 | week 12 after endoscopy
  Number of Participants with Fistula Healing at week 12
Number of Participants with Fistula delay | up to week 18 after endoscopy
  Number of Participants with Fistula delay
Number of Participants with gastric stenosis | up to week 18 after endoscopy
  Number of Participants with gastric stenosis
Measure of length of hospital stay | up to week 18 after endoscopy
  Average total length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sami Hakim, MD, Principal Investigator — CHU Amiens; Jean-Marc Regimbeau, Pr, Principal Investigator — CHU Amiens; Lionel Rebibo, MD, Principal Investigator — Bichat Hospital; Jean-Christophe Duchmann, MD, Principal Investigator — Centre Hospitalier Compiègne; Jonathan Levy, MD, Principal Investigator — Clinique des Cèdres Chât Alliez, Cornebarrieu; Jean-François Bourgaux, MD, Principal Investigator — CHRU Nimes; Ion Donici, MD, Principal Investigator — CHRU Nimes; Vincent Quentin, MD, Principal Investigator — CH Saint Brieux; Fabien Fumex, MD, Principal Investigator — Hopital Jean Mermoz, Lyon; Gaetan Singier, MD, Principal Investigator — Hopital Jean Mermoz, Lyon; Cécile Gomercic, MD, Principal Investigator — CHU NICE; Antonio Iannelli, MD, Principal Investigator — CHU NICE; Claire Blanchard, MD, Principal Investigator — Nantes University Hospital; Timothée Wallenhorst, MD, Principal Investigator — CHU Rennes; Damien Bergeat, MD, Principal Investigator — CHU Rennes; Davide Mazza, MD, Principal Investigator — CH TOULON; Stéphane Koch, MD, Principal Investigator — CHRU Besançon; Nicolas Bouviez, MD, Principal Investigator — CHRU Besançon; Antoine Soprani, MD, Principal Investigator — Clinique Paris-Bercy; Clément Subtil, MD, Principal Investigator — University Hospital, Bordeaux; Ulriikka Chaput, MD, Principal Investigator — Hopital Saint Antoine, Paris; Jérome Rivory, MD, Principal Investigator — Hopital Edouard Herriot - Lyon; Maud Robert, MD, Principal Investigator — Hopital Edouard Herriot - Lyon; Franck Cholet, MD, Principal Investigator — CHU Brest; Jérémie Thereaux, MD, Principal Investigator — CHU Brest; Jean-Christophe Valats, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No